CLINICAL TRIAL: NCT01980537
Title: Stereotaxis and Chronic Total Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Thomas Neunteufl, Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stereotaxis and CTO
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Total Coronary Occlusion

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Stereotaxis (Experimental): Magnetic wire navigation
  Interventions: Procedure: Magnetic wire navigation
- Conventional (Active Comparator): Conventional wire navigation
  Interventions: Procedure: Conventional wire navigation

INTERVENTIONS:
Procedure: Magnetic wire navigation
  Arms: Stereotaxis
Procedure: Conventional wire navigation
  Arms: Conventional

SUMMARY:
Wire-crossing of a chronic total coronary occlusion (CTO) is time-consuming and limited by the amount of contrast agent and time of radiation exposure. Magnetic wire navigation might accelerate wire-crossing by maintaining a coaxial vessel orientation. This study compares magnetic with conventional wire navigation for recanalization of CTOs.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic
* preserved wall motion or viable myocardium
* chronic total occlusion

Exclusion Criteria:

* chronic renal failure
* prior allergic reactions against contrast agent
* hyperthyreosis
* claustrophobia
* pregnancy
* contraindications to aspirin or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
level of contrast medium | 8 hours